CLINICAL TRIAL: NCT03240133
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging, Study to Evaluate the Efficacy, Safety and Tolerability of Single Doses of BCX7353 as an Acute Attack Treatment in Subjects With Hereditary Angioedema
Brief Title: Study of BCX7353 as a Treatment for Attacks of Hereditary Angioedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BCX7353-202
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: HAE; hereditary angioedema; kallikrein inhibitor; plasma kallikrein
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part1: BCX7353 750 mg (Experimental)
  Interventions: Drug: BCX7353
- Part 2: BCX7353 500 mg (Experimental)
  Interventions: Drug: BCX7353
- Part 3: BCX7353 250 mg (Experimental)
  Interventions: Drug: BCX7353
- Parts 1, 2 and 3: placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCX7353 — oral liquid formulation
  Arms: Part 2: BCX7353 500 mg; Part 3: BCX7353 250 mg; Part1: BCX7353 750 mg
Drug: Placebo — oral liquid formulation to match BCX7353
  Arms: Parts 1, 2 and 3: placebo

SUMMARY:
This 3-part study will evaluate the efficacy and safety of an oral kallikrein inhibitor, BCX7353, in the treatment angioedema attacks in subjects with Type I or II hereditary angioedema (HAE). In each study part, subjects will treat 3 attacks with BCX7353 (2 attacks) or placebo (1 attack), in a randomly allocated order. In Part 1, the dose of 750mg will be assessed relative to placebo in up to 36 patients. If this is shown to be effective, then a further 12 patients will be enrolled at a 500mg dose (Part 1), followed by a further 12 (if efficacy still shown) at a dose of 250mg (Part 3) to determine the minimum effective dose of BCX7353 compared to placebo for treating HAE attacks. Efficacy will be determined by subject diary entries completed at pre-defined times post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written, informed consent.
2. A clinical diagnosis of hereditary angioedema Type 1 or Type 2 as documented at any time in the medical records or at the screening visit.
3. Access to and ability to use standard of care acute attack treatment for attacks of HAE.
4. Sexually active women of child-bearing potential and sexually active men must utilize effective contraception.

Exclusion Criteria:

1. Women who are pregnant or breast-feeding.
2. Any clinical condition or medical history that would interfere with the subject's safety or ability to participate in the study.
3. Use of C1INH, androgens or tranexamic acid for prophylaxis of HAE attacks.
4. History of or current alcohol or drug abuse.
5. Infection with hepatitis B, hepatitis C or HIV.
6. Participation in any other investigational drug study currently or within the last 30 days.
7. Positive drugs of abuse screen (unless as used as medical treatment, e.g., with a prescription).
8. An immediate family relationship to either Sponsor employees, the Investigator or employees of the study site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Longhurst, MBBS, PhD, Principal Investigator — Barts & The London NHS Trust
Locations (24):
- Study Center, Graz, Austria
- Study Center, Odense, Denmark
- France (2):
  - Study Center, Grenoble
  - Study Center, Lille
- Germany (2):
  - Study Center, Berlin
  - Study Center, Frankfurt
- Study Center, Budapest, Hungary
- Israel (3):
  - Study Center, Ashkelon
  - Study Center, Tel Aviv
  - Study Center, Tel Litwinsky
- Italy (3):
  - Study Center, Milan
  - Study center, Padua
  - Study Center, Salerno
- Study Center, Skopje, North Macedonia
- Study Center, Krakow, Poland
- Study Center, Târgu Mureş, Romania
- Study Center, Zurich, Switzerland
- United Kingdom (7):
  - Study Center, Birmingham
  - Study Center, Bristol
  - Study Center, Cambridge
  - Study Center, London
  - Study Center, Manchester
  - Study Center, Plymouth
  - Study Center, Southampton

REFERENCES:
- [Derived] Farkas H, Balla Z. A review of berotralstat for the treatment of hereditary angioedema. Expert Rev Clin Immunol. 2023 Feb;19(2):145-153. doi: 10.1080/1744666X.2023.2150611. Epub 2022 Nov 29. PMID 36408587

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: HAE subjects attended a Screening Visit up to 35 days before the baseline visit, for assessment of eligibility to participate in the study.
Groups:
- Part 1: Berotralstat (750 mg) & Placebo Treated HAE Attacks: Each subject treated 3 HAE attacks, 1 with placebo and 2 with 750 mg berotralstat. Placebo vs berotralstat treatment of an HAE attack was assigned by randomization.
- Part 2: Berotralstat (500 mg) & Placebo Treated HAE Attacks: Each subject treated 3 HAE attacks, 1 with placebo and 2 with 500 mg berotralstat. Placebo vs berotralstat treatment of an HAE attack was assigned by randomization.
- Part 3: Berotralstat (250 mg) & Placebo Treated HAE Attacks: Each subject treated 3 HAE attacks, 1 with placebo and 2 with 250 mg berotralstat. Placebo vs berotralstat treatment of an HAE attack was assigned by randomization.
Period: Overall Study
Arm/Group | Part 1: Berotralstat (750 mg) & Placebo Treated HAE Attacks | Part 2: Berotralstat (500 mg) & Placebo Treated HAE Attacks | Part 3: Berotralstat (250 mg) & Placebo Treated HAE Attacks
Started | 33 | 14 | 11
Completed Period 1 | 33 | 14 | 11
Completed Period 2 | 32 | 11 | 11
Completed Period 3 | 30 | 11 | 11
Completed | 30 | 11 | 10
Not Completed | 3 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Rash | 1 | 0 | 0
Not completed — sponsor closure/completion of Part 1 of the study | 1 | 0 | 0
Not completed — Intercurrent illness. | 0 | 1 | 0
Not completed — Sponsor/competent authority/IRB/IEC discontinuation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Berotralstat (750 mg) & Placebo Treated HAE Attacks | Part 2: Berotralstat (500 mg) & Placebo Treated HAE Attacks | Part 3: Berotralstat (250 mg) & Placebo Treated HAE Attacks | Total
Number analyzed (Participants) | 33 | 14 | 11 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 14 | 11 | 57
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.5) | 42.1 (10.5) | 34.9 (10.9) | 41.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 7 | 35
  Male | 16 | 3 | 4 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 33 | 14 | 11 | 58
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 0 | 0 | 1
  Romania | 4 | 0 | 0 | 4
  Hungary | 2 | 0 | 0 | 2
  Denmark | 3 | 0 | 0 | 3
  North Macedonia | 2 | 0 | 0 | 2
  Poland | 2 | 1 | 3 | 6
  Italy | 3 | 4 | 2 | 9
  United Kingdom | 6 | 5 | 2 | 13
  Israel | 4 | 2 | 0 | 6
  France | 1 | 0 | 0 | 1
  Switzerland | 2 | 0 | 0 | 2
  Germany | 3 | 2 | 4 | 9
Adjusted qualifying HAE attack rate [Mean (Standard Deviation); unit: HAE attacks/month] | 3.08 (1.40) | 3.03 (1.23) | 3.23 (1.82) | 3.09 (1.42)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Improved or Stable Composite Visual Analog Scale (VAS) Score
Description: Subjects completed a 3-component VAS on a 100 mm scale for severity of abdominal pain, skin pain and skin swelling associated with the HAE attack, where zero indicated no pain or swelling and 100 mm indicated worst possible pain or swelling. Subjects completed the VAS immediately prior to study drug administration, then at 1, 2, 3, 4, approximately 8 & at 24 hours post-dose. The primary endpoint was the proportion of subject attacks with an improved or stable 3-symptom composite VAS score at 4 hours post dose. The 3-symptom composite was calculated as the average of the VAS scores for abdominal pain, skin pain, and skin swelling. A subject was considered improved or stable if the change from baseline (CFB; time of drug administration) in VAS was ≤ 0.
Time Frame: Mean composite VAS for HAE attack symptoms severity prior to IMP treatment and 4 hours post-dose
Population: The number of participants analyzed in each analysis set corresponds to number of HAE attacks treated with placebo or berotralstat.
Measure: Mean (Standard Deviation); unit: VAS score - millimeters
Units Other Than Participants: HAE Attacks
Groups:
- Part 1: Berotralstat 750 mg - Predose: HAE attack prior to dosing with 750mg berotralstat
- Part 1: Placebo - Pre-dose; Part 2: Placebo - Pre-dose; Part 3: Placebo - Pre-dose: HAE attack prior to dosing with placebo
- Part 1: Berotralstat 750 mg - 4hr Post-dose: HAE attack 4 hr post dosing with 750mg berotralstat
- Part 1: Placebo - 4hr Post-dose; Part 2: Placebo - 4hr Post-dose; Part 3: Placebo - 4hr Post-dose: HAE attack 4 hr post dosing with placebo
- Part 2: Berotralstat 500 mg - Predose: HAE attack prior to dosing with 500mg berotralstat
- Part 2: Berotralstat 500 mg - 4hr Post-dose: HAE attack 4 hr post dosing with 50mg berotralstat
- Part 3: Berotralstat 250 mg - Predose: HAE attack prior to dosing with 250mg berotralstat
- Part 3: Berotralstat 250 mg - 4hr Post-dose: HAE attack 4 hr post dosing with 250mg berotralstat
Arm/Group | Part 1: Berotralstat 750 mg - Predose | Part 1: Placebo - Pre-dose | Part 1: Berotralstat 750 mg - 4hr Post-dose | Part 1: Placebo - 4hr Post-dose | Part 2: Berotralstat 500 mg - Predose | Part 2: Placebo - Pre-dose | Part 2: Berotralstat 500 mg - 4hr Post-dose | Part 2: Placebo - 4hr Post-dose | Part 3: Berotralstat 250 mg - Predose | Part 3: Placebo - Pre-dose | Part 3: Berotralstat 250 mg - 4hr Post-dose | Part 3: Placebo - 4hr Post-dose
Number analyzed (Participants) | 33 | 28 | 33 | 28 | 14 | 9 | 14 | 9 | 11 | 11 | 11 | 11
Number analyzed (HAE Attacks) | 59 | 28 | 59 | 28 | 24 | 9 | 24 | 9 | 21 | 11 | 21 | 11
VAS score - millimeters | 13.96 (9.84) | 15.04 (11.90) | 10.54 (11.39) | 18.42 (14.19) | 17.69 (15.25) | 13.48 (16.11) | 11.31 (15.75) | 9.26 (11.53) | 14.57 (11.78) | 11.33 (10.17) | 10.92 (10.31) | 9.21 (9.67)
Statistical Analysis 1: Comparison: Part 1: Berotralstat 750 mg - Predose vs Part 1: Placebo - Pre-dose vs Part 1: Berotralstat 750 mg - 4hr Post-dose vs Part 1: Placebo - 4hr Post-dose; Change in HAE attack symptoms from pre-dose to 4 hours post-dose was assessed following treatment with either 750mg berotralstat or placebo; Test type: Superiority — Comparisons were performed separately at each time point using a mixed effect linear model including treatment, period and sequence as fixed effects, subject within sequence as a random effect, and predose 3-symptom composite VAS score as a covariate; p = 0.0024, Mixed effect linear model; Difference in Least Square Means = -6.98, 95% CI 2-sided [-11.37 to -2.6]
Statistical Analysis 2: Comparison: Part 2: Berotralstat 500 mg - Predose vs Part 2: Placebo - Pre-dose vs Part 2: Berotralstat 500 mg - 4hr Post-dose vs Part 2: Placebo - 4hr Post-dose; Change in HAE attack symptoms from pre-dose to 4 hours post-dose was assessed following treatment with either 500mg berotralstat or placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6424, Mixed effect linear model; Difference in Least Square Means = -2.1, 95% CI 2-sided [-11.49 to 7.29]
Statistical Analysis 3: Comparison: Part 3: Berotralstat 250 mg - Predose vs Part 3: Placebo - Pre-dose vs Part 3: Berotralstat 250 mg - 4hr Post-dose vs Part 3: Placebo - 4hr Post-dose; Change in HAE attack symptoms from pre-dose to 4 hours post-dose was assessed following treatment with either 250mg berotralstat or placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8283, Mixed effect linear model; Difference in Least Square Means = 0.57, 95% CI 2-sided [-4.9 to 6.03]

2. Primary Outcome: Percentage of Attacks Treated With Standard of Care Acute Attack Medication (SOC-Rx) Through 24 Hours
Description: The proportion of attacks for which subjects took SOC-Rx in the 24 hours following treatment with study drug. HAE Rescue Medications included C1-INH (Berinert, Cinryze, Ruconest) and Firazyr/Icatibant.
Time Frame: 24 hours
Measure: Number; unit: Percentage attacks treated with SOC-Rx
Units Other Than Participants: HAE Attacks
Groups:
- Part 1: Berotralstat 750 mg: HAE attack treated with 750mg berotralstat
- Part 1: Placebo; Part 2: Placebo; Part 3: Placebo: HAE attack treated with placebo
- Part 2: Berotralstat 500 mg: HAE attack treated with 500mg berotralstat
- Part 3: Berotralstat 250 mg: HAE attack treated with 250mg berotralstat
Arm/Group | Part 1: Berotralstat 750 mg | Part 1: Placebo | Part 2: Berotralstat 500 mg | Part 2: Placebo | Part 3: Berotralstat 250 mg | Part 3: Placebo
Number analyzed (Participants) | 33 | 28 | 14 | 9 | 11 | 11
Number analyzed (HAE Attacks) | 59 | 28 | 24 | 9 | 21 | 11
Percentage attacks treated with SOC-Rx | 29.7 | 61.3 | 32.0 | 45.5 | 38.1 | 45.5
Statistical Analysis 1: Comparison: Part 1: Berotralstat 750 mg vs Part 1: Placebo; Analyses were performed using a generalized logistic model including treatment, period and sequence as fixed effects, and subject within sequence as a random effect. The odds of a berotralstat 750 mg-treated-attack requiring SOC-Rx was 0.196 that of a placebo attack; Test type: Superiority; p = 0.0029, logistic mixed effect model; Odds Ratio (OR) = 0.196, 95% CI 2-sided [0.069 to 0.559]
Statistical Analysis 2: Comparison: Part 2: Berotralstat 500 mg vs Part 2: Placebo; Analyses were performed using a generalized logistic model including treatment, period and sequence as fixed effects, and subject within sequence as a random effect. The odds of a berotralstat 500 mg-treated-attack requiring SOC-Rx was 0.472 that of a placebo attack; Test type: Superiority; p = 0.4048, logistic mixed effect model; Odds Ratio (OR) = 0.472, 95% CI 2-sided [0.074 to 2.988]
Statistical Analysis 3: Comparison: Part 3: Berotralstat 250 mg vs Part 3: Placebo; Analyses were performed using a generalized logistic model including treatment, period and sequence as fixed effects, and subject within sequence as a random effect. The odds of a berotralstat 250 mg-treated-attack requiring SOC-Rx was 0.587 that of a placebo attack; Test type: Superiority; p = 0.5984, logistic mixed effect model; Odds Ratio (OR) = 0.587, 95% CI 2-sided [0.073 to 4.733]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from informed consent signature until 16 to 19 days after the 3rd or final HAE attack treated with IMP. As the HAE attack frequency varied between subjects, subject duration of study participation and therefore the duration over which AEs were collected was dependent on attack frequency and therefore variable. The maximum period over which AEs were collected was 281 days.
Description: AEs were assigned to an attack treated with placebo or berotralstat depending on which IMP was used most recently prior to AE onset. HAE attacks and their associated symptoms were not defined as AEs, unless they met the criteria for an SAE.
Groups:
- Part1: Berotralstat 750 mg: Berotralstat : oral liquid formulation
- Part 2: Berotralstat 500 mg; Part 3: Berotralstat 250 mg: Berotralstat: oral liquid formulation
- Parts 1, 2 and 3: Placebo: Placebo: oral liquid formulation to match Berotralstat
Arm/Group | Part1: Berotralstat 750 mg | Part 2: Berotralstat 500 mg | Part 3: Berotralstat 250 mg | Parts 1, 2 and 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/14 | 0/11 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/14 | 0/11 | 1/53
Other Adverse Events (participants affected / at risk) | 12/33 | 8/14 | 7/11 | 17/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1: Berotralstat 750 mg (N=33) | Part 2: Berotralstat 500 mg (N=14) | Part 3: Berotralstat 250 mg (N=11) | Parts 1, 2 and 3: Placebo (N=53)
kidney contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1: Berotralstat 750 mg (N=33) | Part 2: Berotralstat 500 mg (N=14) | Part 3: Berotralstat 250 mg (N=11) | Parts 1, 2 and 3: Placebo (N=53)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In this interim clinical study report (CSR), the VAS change from pre-dose at 4 hours and the proportion of attacks requiring SOC-Rx through the 24 hour post dose were discussed. Assessment of other efficacy endpoints were to be discussed in a final CSR, but this is no longer planned due to a decision to not proceed further with trials of acute treatment of HAE attacks with berotralstat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT03240133/SAP_000.pdf
  • Study Protocol (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT03240133/Prot_001.pdf